CLINICAL TRIAL: NCT01534507
Title: Optimising Measurement of Small and Large Bowel Transit During MRI Scanning and Characterising IBS Subtypes and Their Response to Stress Using MRI (Study 1)
Brief Title: Small and Large Bowel Transit Tests Using MRI (Study 1)
Status: Completed | Type: Observational
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Other Study IDs: 11038; 11/EM/0245 (Study 1) (Other: National Research Ethics Service)
Record Dates: First submitted 2012-02-13; First posted 2012-02-16 (Estimated); Last update posted 2014-08-13 (Estimated); Status verified 2014-08

CONDITIONS: Irritable Bowel Syndrome
MeSH Terms: conditions — Irritable Bowel Syndrome

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Study 1: no samples Study 2: no samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (5):
- Healthy Volunteer 1 (Group 1): For study 1 : Up to 5 healthy volunteers for the initial pilot study and further 21 healthy volunteers for the main study 1
- Group 2 for study 2: Patients with diarrhoea due to irritable bowel syndrome
- Group 3 for study 2: Patients with constipation due to irritable bowel syndrome
- Group 4 for study 2: Patients with mixed bowel habit due to irritable bowel syndrome
- Group 5 for study 2: Healthy volunteer 2: Healthy participants to act as control

SUMMARY:
Irritable bowel syndrome, (IBS) is a common functional disorder of the gut that can be quite disabling to patients. The most common symptoms of IBS are abdominal pain or discomfort along with erratic changes in bowel habit of diarrhoea, constipation or a mixture of the two (referred to as IBS subtypes). Despite much research efforts to further understand the pathophysiology of IBS; as yet no specific biomarkers/definitive measurements have been identified that can be use to aid the diagnosis and reduce the need for unnecessary, unpleasant and expensive tests.

Evidence shows that anxiety plays a part in IBS and can speed up transit time in the small bowel. In this study, the investigators hypothesise that since anxiety is a common feature of IBS, then fast small bowel transit is likely to be found in all subtypes of IBS and the difference in stool frequency and consistency in IBS subgroups are therefore likely to reflect differences in colonic function. The investigator wish to test this by measuring both small and large bowel transit times using Magnetic Resonance Imaging (MRI) and validate the results of the MRI with two methods currently used in clinical practice -The previously validated lactose-C13 Ureide breath test (for small bowel transit) and the standard radio-opaque pellet method to assess the whole gut transit (WGT) time.

DETAILED DESCRIPTION:
The investigator has 2 main parts in this study i.e. Study 1 and Study 2.

As part of study 1, the investigator would like to recruit up to 5 healthy volunteers as a pilot study to optimise measurement and analysis of the Lactose-C13 Ureide breath test along with MRI scannings at regular intervals.

Following from this, the investigator would like assess the feasibility and reproducibility of using MRI imaging to assess gastrointestinal transit. The investigator would like to recruit 21 healthy volunteers to measure orocaecal transit time (OCTT) and whole gut transit(WGT)using the conventional method of Lactose-C13 Ureide breath test for OCTT and the Metcalf method using standard radio-opaque pellet method for WGT and compare them will MRI imaging. Once this has been analysed and the best method for each OCTT and WGT have been decided, these methods would be applied in Study 2.

In study 2, the investigator would like to recruit 30 healthy volunteers, 30 patients with diarrhoea predominantly Irritable Bowel Syndrome, 30 patients with constipation predominantly Irritable Bowel Syndrome and 30 patients with Mixed irritable Bowel Syndrome. The best methods from study 1 for OCTT and WGT will be applied here to assess gastrointestinal transit on these subjects. Based on the first study, the best method to assess OCTT is the Lactose-C13 Ureide breath test and for the WGT, the best method is the MRI marker capsules. Participants will need to fill in questionnaires to assess their stress levels and to fill in symptom questionnaires during the study day.

ELIGIBILITY:
Study 1

Inclusion Criteria

* 26 healthy volunteer
* Age 18-75 years old
* Non-smoker
* Able to give informed consent

Exclusion Criteria

* Lactose intolerant
* Any history of gastrointestinal surgery on the small bowel (excluding appendicectomy)
* Pregnancy
* contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury alcohol dependence
* serious concomitant illness as judged by the investigators
* use of drugs known to alter GI motility including opiates, anti-depressants, selective serotonin reuptake inhibitors, tricyclic antidepressants, monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists during or in the 2 weeks prior to the test
* inability to lie flat or exceed scanner limits of weight >120kg or abdominal circumference >99cm ; BMI <18 and >30 kg/m2
* Poor command of English language
* Participation of any medical trials for the past 3 months

Study 2:

120 participants consisting of: 30 patients with diarrhoea predominant IBS according to Rome III criteria 30 patients with constipation predominant IBS according to Rome III criteria 30 patients with mixed type IBS according to Rome III criteria 30 healthy volunteers age and sex matched controls

Inclusion criteria

* Meet the Rome III criteria and the IBS subtypes
* Age 18-75 years old
* Able to give informed consent
* Subjects will undergo a limited screening medical. They will also complete a MRI - safety questionnaire and be given an information sheet
* Able to give informed consent
* Subjects will undergo screening medical questionnaire. They will also complete a MRI safety questionnaire and be given an information sheet

Exclusion Criteria

* Any history of gastrointestinal surgery on the small bowel (excluding appendicectomy)
* Pregnancy
* contraindications for MRI scanning i.e. metallic implants, pacemakers, history of metallic foreign body in eye(s) and penetrating eye injury
* alcohol dependence
* serious concomitant illness as judged by the investigators
* use of drugs known to alter GI motility including opiates, , monoamine oxidase inhibitors, phenothiazines, benzodiazepines, calcium channel antagonists during or in the 2 weeks prior to the test
* Selective serotonin reuptake inhibitors or low dose tricyclic antidepressants will be recorded but will not be an exclusion
* No recent antibiotic treatment past 2 weeks
* inability to lie flat or exceed scanner limits of weight >120kg or abdominal circumference >99cm; BMI <18 and >30 kg/m2
* Poor command of English language
* Participation of any medical trials for the past 3 months

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy volunteers will be selected via poster advertisement Participants with Irritable Bowel Syndrome will be selected from the gastroenterology clinics /poster advertisement
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2011-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Study 1:Correlation between mean orocaecal transit time as assessed by MRI and lactose C13-ureide | 9 hours
  MRI:Orocaecal transit time (OCTT) can be measured by the first scan showing arrival of the head of a meal in the ascending colon Lactose C13-Ureide breath test:Orocaecal transit time will be taken as the time at which a significant increase from background in breath 13C was seen.
Study 1: Correlation between colonic transit as assessed by from the geometric centre of the PTFE capsule at time 24 and 48 hours and Metcalf Radio-opaque marker method | 72 hours
  Colonic transit using MRI will be measure by assessing the geometric centre position in colon/small bowel.
  Whole gut transit time using the Metcalf method of Radio-opaque Marker method would be estimated by counting the number of pellets remaining in the colon in an abdominal x-ray taken in day 4 * 1.2
Study 2: Fasting small bowel water content | 1 hour
  Fasting small bowel water content (SBWC) in the 3 subgroups of Irritable Bowel Syndrome (IBS) compared to healthy controls

SECONDARY OUTCOMES:
Study 1:To assess reproducibility of the using MRI for orocaecal transit time and colonic transit time | 21 days
  In study 1, the orocaecal transit time and colonic transit time would be repeated twice with a week break in between to assess reproducibility of the MRI.
Study 2: Orocaecal transit time using lactose C13-ureide | 9 hours
  Orocaecal transit time in the 3 subgroups of IBS versus healthy control using the best method from study 1 which is the lactose C13-Ureide breath test
Study 2: Area under the curve (AUC) post prandial SBWC | 9 hours
Study 2: Ascending colon water content (ACWC) and colonic water index (CWI) | 9 hours
Study 2: Colonic volumes both fasting and post prandial (divided into ascending transverse and descending colon) | 9 hours
Study 2: Whole gut transit time assess by MRI marker capsule from study 1 | 24 hours
  The best method to assess the whole gut transit time based on study 1 was the use of the MRI marker capsule at time 24hours
Study 2: Correlation between the Hospital Anxiety & Depression Scale (HADS) and other measures of anxiety and stress score and (a) Oro-caecal transit time and (b)whoe gut transit time | 9hours

CONTACTS AND LOCATIONS:
Overall Officials: Robin Spiller, MD FRCP, Study Director — University of Nottingham; Ching Lam, MBchB MRCP, Principal Investigator — University of Nottingham
Locations (1):
- University of Nottingham, Nottingham, Notts, United Kingdom

REFERENCES:
- [Background] Metcalf AM, Phillips SF, Zinsmeister AR, MacCarty RL, Beart RW, Wolff BG. Simplified assessment of segmental colonic transit. Gastroenterology. 1987 Jan;92(1):40-7. doi: 10.1016/0016-5085(87)90837-7. PMID 3023168
- [Result] Chaddock G, Lam C, Hoad CL, Costigan C, Cox EF, Placidi E, Thexton I, Wright J, Blackshaw PE, Perkins AC, Marciani L, Gowland PA, Spiller RC. Novel MRI tests of orocecal transit time and whole gut transit time: studies in normal subjects. Neurogastroenterol Motil. 2014 Feb;26(2):205-14. doi: 10.1111/nmo.12249. Epub 2013 Oct 25. PMID 24165044